CLINICAL TRIAL: NCT04294888
Title: TMS in Preclinical and Prodromal AD: Modulation of Brain Networks and Memory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jessica A. Collins, PhD, Instructor, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019P003445
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Aging
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Participants will each undergo, in a crossover, within-subject design, two blocks of rTMS: active and SHAM.The order of active and SHAM blocks will be counterbalanced across subjects.
Who Masked: Participant
Masking Description: All participants will undergo SHAM stimulation as a control condition. They will be blinded as to whether they are receiving active or SHAM stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active stimulation (Experimental): Active rTMS will be administered with a MagPro X100 stimulator (MagVenture, Denmark), using a 70 mm figure-of-eight liquid cooled coil capable of doing active or sham stimulation (e.g. the Cool B70 coil or the Cool B65 A/P coil). Active rTMS will be delivered at 80% of a patient's active motor threshold. rTMS will be administered in an excitatory iTBS pattern. Stimulation parameters will remain well within established safety guidelines (Rossi et al. 2009).
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)
- Sham stimulation (Sham Comparator): SHAM stimulation will also be administered with a MagPro X100 stimulator (MagVenture, Denmark), using a 70 mm figure-of-eight liquid cooled coil capable of doing active or sham stimulation (e.g. the Cool B70 coil or the Cool B65 A/P coil). SHAM rTMS will be delivered at 80% of a patient's active motor threshold. SHAM stimulation will be delivered to the exact same cortical targets as active rTMS. While no electromagnetic stimulation will be delivered during SHAM, the sounds will approximate active stimulation and skin electrodes will approximate the sensation of active rTMS. Inclusion of a sham condition in this protocol is critical to measure whether or not the stimulation is improving memory performance, or whether practice effects or other non-specific effects are responsible for any changes in memory which may be observed.
  Interventions: Device: repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation (rTMS) — rTMS is a method to focally and reversibly stimulate a pre-specified cortical target. rTMS works through the principle of electromagnetic induction.

SUMMARY:
The purpose of this study is to assess the effects of non-invasive brain stimulation on memory in cognitively unimpaired older adults and in patients amnestic mild cognitive impairment (aMCI) due to Alzheimer's disease (AD). This study will use repetitive Transcranial Magnetic Stimulation (rTMS) to stimulate nodes of the Default Mode Network (DMN)- which is thought to support episodic memory and to be affected by Alzheimer's pathology.

We will use functional connectivity MRI (fcMRI) to assess changes in functional network architecture following the stimulation. We will also assess putative cognitive improvements resulting from the stimulation by in-depth memory testing.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 60-85
2. All participants will be native English speakers
3. Willing and able to consent to the protocol and undergo imaging and neuropsychological testing at the specified time points
4. Participants with aMCI will be asked to bring a study partner to all visits
5. Only patients with very mild or mild cognitive impairment (CDR 0.5 or CDR 1) will be included in the prodromal AD cohort

Exclusion Criteria:

1. History of head trauma involving loss of consciousness or alteration in consciousness
2. Another major neurologic or psychiatric condition
3. Known presence of a structural brain lesion (e.g. tumor, cortical infarct)
4. Any contraindication to MRI, such as presence of pacemakers, aneurysm clips, artificial heart valves, ear implants, metal fragments, or foreign objects in the eyes, skin, or body
5. Longstanding premorbid history (i.e. longer than 10 years) of alcohol or substance abuse with continuous abuse up to and including the time that the symptoms leading to clinical presentation developed
6. Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the study protocol.
7. Unwilling to return for follow-up, undergo neuropsychological testing, TMS, and MR imaging

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Paired Associative Face Name Memory Test | up to 5 weeks
  A test of memory for face-name associations

SECONDARY OUTCOMES:
Changes in intrinsic functional connectivity | up to 5 weeks
  Changes in region-to-region functional connectivity within the stimulated network will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Massachuetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with researchers outside of this protocol.